CLINICAL TRIAL: NCT01187056
Title: The RISAP-study: a Complex Intervention in Risk Communication and Shared Decision-making in General Practice
Acronym: RISAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007-41-1446
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2012-10

CONDITIONS: High Cholesterol; Cardiovascular Disease
Keywords: Shared decision-making; Risk information; Decision aids
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training, decision making (Experimental): General practitioners receive training in shared decision-making and risk communication, and use their newly acquired skills in real-life consultations with 7 patients with high cholesterol.
  Interventions: Behavioral: Training programme
- Training, usual practice (Active Comparator): The control group GPs will receive 2 hours of training in the primary care guideline for prevention of cardiovascular disease
  Interventions: Behavioral: Training programme

INTERVENTIONS:
Behavioral: Training programme — 2 x 2 hours of training (workshops)
  Other Names: decision making, decision aids

SUMMARY:
General practitioners (GPs) and patients find it difficult to talk about risk of future disease, especially when patients have asymptomatic conditions, and treatment options are unlikely to cause immediate perceptible improvements in well-being. Further studies in risk communication for disease prevention are needed, as are studies about risk communication training for GPs. Aim: 1) to systematically develop, describe and evaluate a complex intervention comprising a training programme for GPs in risk communication and shared decision-making, 2) to evaluate the effect of the training programme on real-life consultations between GPs and patients with high cholesterol levels, and 3) to evaluate patients' reactions during and after the consultations. Hypothesis: 1) patients have better adherence to chosen treatment.

The effect of the complex intervention, based around a training programme, will be evaluated in a cluster-randomised controlled trial with an intervention group and an active control group with 40 GPs and 280 patients in each group.

The GPs receive a questionnaire at baseline and after 6 months about their attitudes towards risk communication and cholesterol-reducing medication. After each consultation with a participating high cholesterol-patient, the GPs will complete a questionnaire about decision satisfaction.

The patients will receive a questionnaire at baseline and after 3 and 6 months. It includes questions about adherence to chosen treatment, self-rated health, patient enablement, and risk communication and decision-making effectiveness. Prescriptions, contacts to the health services, and cholesterol level will be drawn from the register of the National Health Service of Denmark at baseline and at 6 months.

In both intervention group and active control group, 12 consultations will be observed and tape-recorded. The consultations will be divided between 4 GPs with each 3 patients. The patients from these 24 consultations will be interviewed immediately after the consultation and re-interviewed after 6 months.Eight purposefully selected GPs from the intervention group will be interviewed in a focus group 6 months after participation in the training programme. The process and context of the RISAP-study will be investigated in detail using an action research approach, in order to describe and analyse research choices, adaptation of intervention model to the specific context, and GPs' and patients' reactions to trial participation.

ELIGIBILITY:
Inclusion Criteria:

- GPs in Region Central and Region North, Denmark, are invited to the study.

Patients are at least 18 years old, and have high cholesterol corresponding to a recommendation for cholesterol-reducing medication according to Danish clinical guideline for general practice. The patients are recruited after their high cholesterol has been detected and when treatment options are to be discussed.

Exclusion Criteria:

- Patients with CVD or DM are excluded from the study, as are patients already receiving cholesterol-reducing medication and patients unable to speak and read Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary patient outcome is adherence to treatment choice. | 2010-08-01 - 2011-04-01

SECONDARY OUTCOMES:
satisfaction with decision. | 2010-08-01 - 2011-04-01
self-rated health | 2010-08-01 - 2011-04-01
anxiety | 2010-08-01 - 2011-04-01
enablement | 2010-08-01 - 2011-04-01
satisfaction with communication, | 2010-08-01 - 2011-04-01
satisfaction and confidence in decision | 2010-08-01 - 2011-04-01
number of contacts to health services | 2010-08-01 - 2011-04-01

CONTACTS AND LOCATIONS:
Overall Officials: Janus L Thomsen, MD, PhD, Principal Investigator — University of Aarhus

REFERENCES:
- [Derived] Kirkegaard P, Edwards A, Risor MB, Thomsen JL. Risk of cardiovascular disease? A qualitative study of risk interpretation among patients with high cholesterol. BMC Fam Pract. 2013 Sep 16;14:137. doi: 10.1186/1471-2296-14-137. PMID 24040920
- [Derived] Kirkegaard P, Risor MB, Edwards A, Junge AG, Thomsen JL. Speaking of risk, managing uncertainty: decision-making about cholesterol-reducing treatment in general practice. Qual Prim Care. 2012;20(4):245-52. PMID 23113909
- [Derived] Kirkegaard P, Edwards AG, Hansen B, Hansen MD, Jensen MS, Lauritzen T, Risoer MB, Thomsen JL. The RISAP-study: a complex intervention in risk communication and shared decision-making in general practice. BMC Fam Pract. 2010 Sep 22;11:70. doi: 10.1186/1471-2296-11-70. PMID 20860820